CLINICAL TRIAL: NCT01842438
Title: Psychosexual Support Following Prostate Cancer Surgery: Feasibility and Outcomes of a Couple-based Intervention
Brief Title: A Couple Support Intervention for Prostate Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Stirling (Other)
Collaborators: Prostate Cancer UK (Other)
Responsible Party: Principal Investigator, Prof Liz Forbat, Reader, University of Stirling
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 03979
Record Dates: First submitted 2013-04-24; First posted 2013-04-29 (Estimated); Results first posted 2016-06-22 (Estimated); Last update posted 2017-06-05 (Actual); Status verified 2017-05

CONDITIONS: Prostate Cancer
Keywords: Sexual Dysfunctions, Psychological
MeSH Terms: conditions — Prostatic Neoplasms; Sexual Dysfunctions, Psychological

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Behavioral: psychosexual intervention (Experimental): 6-sessions of couple support focused on relationships and psychosexual functioning
  Interventions: Behavioral: Behavioral: psychosexual intervention
- Control (No Intervention): This group will not receive the intervention during the life-span of the project

INTERVENTIONS:
Behavioral: Behavioral: psychosexual intervention — 6 session manualised intervention, This manual-based family-relational-psychosexual support was based on systemic principles combined with techniques from sex therapy, i.e. sensate focus. The manual offered an intermediate level of specificity, enabling practitioners to use their own therapeutic style and take some lead from the couple while meeting the objectives of the intervention. Specialist training in delivery of the intervention was provided to practitioners holding accredited counselling or psychotherapy qualifications. Practitioners engaged in routine clinical supervision with one additional team supervision session offered by one of the practitioners
  Arms: Behavioral: psychosexual intervention

SUMMARY:
Even with careful prostate surgery, men find it difficult to have an erection. Our previous research shows that couples are not often supported to cope with the effects of surgery on their sexual relationships. In this study, the investigators will design a way of supporting couples, and test how well it works.

The investigators will decide what the support should include (e.g. duration, frequency and timing of the support). The investigators will do this by looking at available literature on the subject.

The investigators will recruit 68 couples to the study, half will receive standard care and the other half will be invited to attend six sessions of psychosexual support with specially trained professionals (trained by men affected by prostate conditions and a cancer/couple support specialist). Before and after the support, men and their partners will be asked to complete questionnaires which measure quality-of-life, emotional needs, and their relationship. The investigators will ask the couples to fill out the questionnaires again six-months later to see if the support has long-term benefits. At the end of the study the investigators will also interview 10 couples to find out their views of the support, and another 10 couples about standard treatment.

When the investigators have tested this support, they expect to see men and their partners tell us that their quality of life has improved, and they have higher satisfaction with their relationship. The investigators will calculate the overall cost of providing this support, and the benefits it has on reducing the need for other health-care services (like General Practice use).

DETAILED DESCRIPTION:
Scientific abstract

Evidence shows significant unmet psychosexual needs for couples affected by prostate cancer. Studies have identified the contribution that psychosocial interventions could have for couples, e.g. strengthening healthy adaptation and better communication, developing coping skills for distressed couples, and facilitating healthy spousal communication to address the sexual rehabilitation needs.

This is a feasibility study with a built-in pilot, which will examine the acceptability, feasibility and outcomes of a psychosexual intervention to support couples, drawing on the Medical Research Council complex intervention framework.

The intervention will be developed from the extant and our pilot work. Men in outpatient surgical follow-up clinics will be screened using EPIC, and recruited if scoring under the clinical threshold for potency. 68 couples will be randomised to two arms, one receiving six sessions of couple-support from specially trained counsellors and the others receiving standard care. The primary outcome measure is health-related quality-of-life. Pre, post and 6-month follow-up outcomes will be measured in both individual (quality of life; anxiety/depression) and in relational terms (relationship between couples). An economic analysis will identify population costs.

ELIGIBILITY:
Inclusion Criteria:

* Score of ≤60 on EPIC (a signal of potency) (EPIC is the Expanded Prostate Cancer Index Composite)
* >11 weeks post-operative for Prostate Cancer (PCa) (to recruit people who have recovered from the immediate effects from surgery and begun to regain some functioning. Follow-ups are held at 6weeks, 12weeks, 6months from surgery, until no further follow-up is required).
* Has a partner

Exclusion Criteria:

* Does not have a partner (this is a couple intervention, the study can therefore only include men with a partner).
* Prognosis of ≤1year (Most men who have had recent surgery will have a good prognosis, consequently it is unlikely that many men will be excluded by this criteria.)
* Unable to provide informed consent.
* Residing in Dumfries and Galloway. The recruiting clinic sees patients from a wide catchment area. However to prevent excess burden on participants traveling to the intervention site in Edinburgh, the investigators will exclude those living in Dumfries and Galloway.
* >2 years from surgery (since long term adaptation will have commenced).
* Unable to communicate in English (this is a feasibility trial, if the study moves to a full scale trial in future then it will seek to include couples and interpreters/translators).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2012-10; Primary Completion 2015-07 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Liz Forbat, PhD, Principal Investigator — University of Stirling
Locations (1):
- Western General Hospital, Edinburgh, Lothian, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Consent was not gained for data sharing in this manner

REFERENCES:
- [Derived] Robertson JM, Molloy GJ, Bollina PR, Kelly DM, McNeill SA, Forbat L. Exploring the feasibility and acceptability of couple-based psychosexual support following prostate cancer surgery: study protocol for a pilot randomised controlled trial. Trials. 2014 May 24;15:183. doi: 10.1186/1745-6215-15-183. PMID 24886676

RESULTS

PARTICIPANT FLOW:
Groups:
- Behavioral: Psychosexual Intervention: 6-sessions of couple support focused on relationships and psychosexual functioning
  Behavioral: psychosexual intervention
Period: T1: Immediately After the Intervention
Arm/Group | Behavioral: Psychosexual Intervention | Control
Started | 42 | 44
Completed | 36 | 36
Not Completed | 6 | 8
Not completed — Withdrawal by Subject | 6 | 8
Period: T2: 6month Follow-up
Arm/Group | Behavioral: Psychosexual Intervention | Control
Started | 36 | 36
Completed | 32 | 32
Not Completed | 4 | 4
Not completed — Withdrawal by Subject | 4 | 3
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Behavioral: Psychosexual Intervention | Control | Total
Number analyzed (Participants) | 42 | 44 | 86
Age, Continuous [Mean (Standard Deviation); unit: years] — Data was collected only for patient participants (all of whom were male)
  years | 64.15 (6.885) | 63.27 (8.800) | 63.72 (7.772)
Sex/Gender, Customized [Number; unit: participants]
  Male | 22 | 22 | 44
  Female | 20 | 22 | 42
Region of Enrollment [Number; unit: participants]
  United Kingdom | 42 | 44 | 86
EPIC sexual bother subscale (prostate-specific quality of life) [Mean (Full Range); unit: units on a scale] — Higher scores indicate better outcomes (better functioning; less bother). This measure was only completed by patients (all of whom were male).
  units on a scale | 24.11 [0 to 62.5] | 20.45 [0 to 62.5] | 22.28 [0 to 62.5]

OUTCOME MEASURES:

1. Primary Outcome: EPIC (Expanded Prostate Cancer Index Composite), Sexual Bother Subscale
Description: EPIC is a quality of life tool used in prostate cancer studies, focused on physical and sexual outcomes. It is validated with population norms. We used the sexual bother sub-scale as the primary outcome measure; score range 0-400. A higher score indicates better function/better outcome.
Time Frame: Basline (T0), immediate post-intervention (T1) and 6 Months (T2)
Population: Primary outcome was at T1, sample size at T1, n=21 intervention, n=22 control. Sample size at T2, n=13 intervention, n=14 control At T1 (immediate follow-up) 3 intervention patients had withdrawn and 4 control patients had withdrawn. The scale was completed only by patients (all of whom were men, by as study focused on prostate cancer).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Behavioral: Psychosexual Intervention | Control
Number analyzed (Participants) | 21 | 22
units on a scale
  Patients T0 | 24.11 (20.38) | 20.45 (21.14)
  Patients T1: number analyzed (Participants) | 18 | 18
  Patients T1 | 44.092 (30.42833) | 26.3889 (23.243)
  Patients T2: number analyzed (Participants) | 14 | 16
  Patients T2 | 30.77 (32.12) | 29.91 (31.41)

2. Secondary Outcome: HADS (Hospital Anxiety and Depression Scale)
Description: The HADS has two scales: one anxiety and one depression. It is validated with population norms. Results are presented for T2 (6 month follow-up) and split by Patient, Partner and again by Intervention, Control.
  Responses are scored on a scale of 0-3 (3 indicates higher symptom frequencies. Scores for each subscale (anxiety and depression) range from 0 to 21 with scores categorized as follows: normal 0-7, mild 8-10, moderate 11-14, and severe 15-21. Scores for the entire scale (emotional distress) range from 0 to 42, with higher scores indicating more distress.
Time Frame: Basline (T0), immediate post-intervention (T1) and 6 Months (T2)
Population: Data received at each time-point was T0: intervention, T1: immediately after intervention; T2 6months post intervention.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Behavioral: Psychosexual Intervention PATIENTS: 6-sessions of couple support focused on relationships and psychosexual functioning
  Behavioral: psychosexual intervention
  This data is patients-only (all males)
- Intervention: Partners: This group received the intervention during the life-span of the project. Partners only.
- Control: Patient Group: Did not receive the intervention. All males
- Control: Partners: Did not receive the intervention; mostly females, but one male as there was one same-sex couple participating.
Arm/Group | Behavioral: Psychosexual Intervention PATIENTS | Intervention: Partners | Control: Patient Group | Control: Partners
Number analyzed (Participants) | 21 | 21 | 22 | 22
units on a scale
  HADS total (T0) | 10.67 (6.87) | 11.14 (5.842) | 9.77 (6.406) | 8.55 (6.69)
  Anxiety subscale only (T0) | 6.24 (4.146) | 7.71 (3.59) | 6.32 (4.12) | 5.82 (4.57)
  Depression subscale only (T0) | 4.43 (3.56) | 3.43 (2.84) | 3.45 (2.72) | 2.73 (2.95)
  HADS total (T1): number analyzed (Participants) | 18 | 18 | 22 | 22
  HADS total (T1) | 7.22 (5.92) | 6.98 (4.95) | 8.94 (6.20) | 8.72 (6.58)
  Anxiety subscale only (T1): number analyzed (Participants) | 18 | 18 | 18 | 18
  Anxiety subscale only (T1) | 4.06 (3.42) | 5.17 (3.60) | 5.72 (4.11) | 6.33 (4.99)
  Depression subscale only (T1): number analyzed (Participants) | 18 | 18 | 18 | 18
  Depression subscale only (T1) | 3.17 (3.22) | 1.72 (2.02) | 3.22 (2.46) | 2.39 (2.63)
  HADS total (T2): number analyzed (Participants) | 14 | 14 | 16 | 16
  HADS total (T2) | 7.93 (5.980) | 5.57 (4.586) | 10.44 (7.624) | 9.19 (7.250)
  Anxiety subscale only (T2) | 4.29 (3.197) | 4.07 (2.674) | 6.69 (5.885) | 6.31 (5.510)
  Depression subscale only (T2): number analyzed (Participants) | 14 | 14 | 16 | 16
  Depression subscale only (T2) | 3.64 (3.365) | 1.5 (3.082) | 3.75 (2.646) | 2.88 (3.324)

3. Secondary Outcome: SCORE15 (Systemic Core Outcome Measure)
Description: SCORE15 is an index of Family Function and Change, with 15 items. The potential range of scores is 15 to 75, with a lower score indicating higher family functioning. Total scores are reported in the data below.
Time Frame: Basline (T0), immediate post-intervention (T1) and 6 Months (T2)
Population: Data received at each time-point was T0: intervention 42, control: 43; T1: intervention 36, control 36; T2 (as above) intervention 28, control 32
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Behavioral: Psychosexual Intervention | Control
Number analyzed (Participants) | 28 | 32
units on a scale
  Patients T0 | 22.14 (5.825) | 27.52 (10.934)
  Partners T0 | 24.38 (9.357) | 25.82 (7.986)
  Patients T1 | 22.31 (7.181) | 27.50 (11.377)
  Partners T1 | 22.67 (6.221) | 22.11 (6.807)
  Patients T2 | 25.14 (9.550) | 29.25 (12.402)
  Partners T2 | 21.64 (6.868) | 24.69 (10.423)

ADVERSE EVENTS:
Time Frame: Participants were followed for the duration of the trial, from return of consent form to completion of the T2 measures (6months following the end of the intervention)
Arm/Group | Behavioral: Psychosexual Intervention | Control
Serious Adverse Events (participants affected / at risk) | 0/42 | 0/44
Other Adverse Events (participants affected / at risk) | 0/42 | 0/44

LIMITATIONS AND CAVEATS:
Under-recruitment means the study is not powered (though the study was designed as a pilot, so not hypothesis testing).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes